CLINICAL TRIAL: NCT00990873
Title: A Validation of the 64-Gene Signature Using Affymetrix-HG_U133A Array in Stage I NSCLC From the CALGB Lung Cancer Study (140202)
Brief Title: Study of Tissue Samples From Patients With Stage I Non-Small Cell Lung Cancer Enrolled on Research Study CALGB-140202
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150803; CALGB-150803; CDR0000649826 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissues and blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tissue samples from patients with stage I non-small cell lung cancer enrolled on research study CALGB-140202.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the 64-gene signature can accurately predict the prognosis for survival of patients with stage I non-small cell lung cancer (NSCLC).

OUTLINE: RNA is purified from tissue samples obtained by the CALGB Lung Cancer Study (CALGB-140202). The RNA samples are used for gene expression analysis using the 64-gene signature and an Affymetrix-HG_U133A array. Reverse-transcriptase PCR may also be performed on selected samples.

ELIGIBILITY:
1. Registration to CALGB 140202
2. Institutional Review Board (IRB) review and approval at the institutions where the laboratory work will be performed is required
3. Informed Consent: The CALGB does not require that a separate consent form be signed for this study

   * The subject population to be studied in this protocol includes patients selected from CALGB 140202. All such patients have signed a written informed consent document meeting all federal, state and institutional guidelines as part of entry into that trial.
   * All samples to be studied were obtained and stored as part of CALGB 140202. The material and data obtained from the patient's protocol record will be used to obtain appropriate clinical information. In no instance will the patient be contacted directly.
   * There should be no physical, psychological, social or legal risks associated with this study. No invasive procedures are recommended or requested.
   * All appropriate and necessary procedures will be utilized to maintain confidentiality. All patients who have had samples submitted for analysis will have their CALGB study number used to identify specimens.
   * This study does not require direct patient contact and no specific risk or benefits to individuals involved in the trial are anticipated. It is likely however, that the information gained will substantially help similar patients in the future.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage I non-small cell lung cancer and previously enrolled on CALGB 140202.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Overall survival, defined as the time from surgery to death of any cause | Up to 5 years

SECONDARY OUTCOMES:
Disease-free survival, defined as time from surgery to any recurrence (local or regional), second primary tumor, distant metastasis, or death of any cause | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ming You, MD, Study Chair — Washington University Siteman Cancer Center